CLINICAL TRIAL: NCT02913144
Title: Implication of a Coronary Calcium Screening Examination, Incidence of Cardiovascular Events and Progression of Coronary Artery Calcium Over up to 7 Year of Follow-up in a Danish Middle-aged General Population
Brief Title: 7 Year Follow-up Study of the DanRisk Population
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Mette Hjortdal Grønhøj, M.D, Odense University Hospital
Other Study IDs: 13/31879
Record Dates: First submitted 2016-07-19; First posted 2016-09-23 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-07

CONDITIONS: Cardiovascular Disease; Coronary Artery Calcification; Atherosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Biospecimen Retention: Samples Without DNA — a biobank consisting of plasma and serum was established in 2009 and also in 2014-15.
Oversight: Data Monitoring Committee: No

SUMMARY:
OBJECTIVES: To investigate the incidence of cardiovascular events as well as progression of coronary artery calcium (CAC) in healthy middle-aged subjects over a period of 7 years, and the relation to traditional as well as new cardiovascular risk factors.

METHODS: The Danrisk cohort was established in 2009-2010 based on random retrieval from the Danish national civil registry (N=1825). Initially, distribution of gender, area of residence and year of birth (1949 or 1959) were equal among the 4 involved centres (OUH, Svendborg, Vejle and Esbjerg). A total of 1257 subjects (69%) accepted the invitation to undergo cardiovascular risk evaluation including non-contrast enhanced cardiac CT-scan for CAC estimation, and a total of 1227 subjects were found free of cardiovascular disease (CVD) and diabetes (DM), and was included in the study back then.

In 2014-2015 the DanRisk cohort was invited to a 5 year follow-up examination. The investigators examined a total of 1031 subjects (82%) in the investigators 4 regional centres. The follow-up examination included general health evaluation and estimation of CAC by non-contrast enhanced cardiac CT-scan. Information of death, cardiovascular events and medication usage was obtained from the Danish national patient register, the Danish register of causes of death and the Danish national database of reimbursed prescriptions in 2016.

ELIGIBILITY:
Inclusion Criteria:

* Born in either 1949 or 1959
* Residence in/near one of the regional centres (Esbjerg, Svendborg, Vejle, Odense).

Exclusion Criteria:

* Known cardiovascular disease

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Danrisk cohort was established in 2009-2010 based on random retrieval from the Danish national civil registry (N=1825). Initially, distribution of gender, area of residence and year of birth (1949 or 1959) were equal among the 4 involved centres (OUH, Svendborg, Vejle and Esbjerg). A total of 1257 subjects (69%) accepted the invitation to undergo cardiovascular risk evaluation including non-contrast enhanced cardiac CT-scan for CAC estimation, and a total of 1227 subjects were found free of CVD and DM, and was included in the study back then.
  In 2014-2015 the DanRisk cohort was invited to a 5 year re-examination. The investigators examined a total of 1031 subjects (82%) in the investigators 4 regional centres.
Sampling Method: Non-Probability Sample
Enrollment: 1257 (Actual)
Dates: Start 2014-05; Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Incident CV event | 6.5 years

SECONDARY OUTCOMES:
CAC Progression | 5 years

IPD SHARING:
Plan to Share IPD: Undecided